CLINICAL TRIAL: NCT00109473
Title: A Phase II Randomized Trial of Growth Hormone Therapy in Pediatric Crohn's Disease
Brief Title: Trial of Growth Hormone Therapy in Pediatric Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHMC IRB #: 04-12-06; IND # 71,344 (Other: FDA)
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Crohn's Disease
Keywords: Pediatric Crohn's disease; Pediatric; Crohn's Disease
MeSH Terms: conditions — Crohn Disease; Pediatric Crohn's disease | interventions — Growth Hormone; Prednisone; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth Hormone plus cortecosteroid (Experimental): Growth Hormone (nutropin AQ 0.075 mg/kg/day subcutaneously daily)
  Interventions: Drug: growth hormone
- Cortecosteroids alone (Active Comparator): Cortecosteroid therapy as prescribed by the referring gastroenterologist
  Interventions: Drug: cortecosteroid

INTERVENTIONS:
Drug: growth hormone — Nutropin AQ 0.075mg/kg/day subcutaneously daily
  Other Names: Nutropin AQ
  Arms: Growth Hormone plus cortecosteroid
Drug: cortecosteroid — As prescribed by the referring gastroenterologist
  Other Names: Prednisone, Entocort
  Arms: Cortecosteroids alone

SUMMARY:
The purpose of this study is to determine whether taking a growth hormone (GH) drug called somatropin causes the intestine of a person with Crohn's Disease (CD) to heal faster when compared to a person with Crohn's Disease that does not receive growth hormone drug.

DETAILED DESCRIPTION:
The optimal treatment goals in childhood CD include: 1) clinical remission in conjunction with mucosal healing and 2) restoration of normal growth and development. Current therapy in most cases includes induction of remission with corticosteroids followed by maintenance of remission with 6-mercaptopurine (6-MP) or mesalamine. With this approach, the goals of achieving mucosal healing with normalization of growth are not achieved in a significant number of children. GH therapy is now used in several chronic childhood diseases which are complicated by growth failure despite adequate GH secretion. These include chronic renal failure (CRF), juvenile rheumatoid arthritis (JRA), and Turner's syndrome. However, despite a comparable frequency and magnitude of permanent growth failure, the efficacy of GH therapy in this respect has not yet been determined in a controlled trial for CD. Moreover, whether GH therapy may also directly reduce disease activity and promote intestinal healing is not known. This represents a significant clinically unmet need in this patient population. Therefore, new therapeutic approaches are needed to both improve final adult height and enhance intestinal mucosal healing in children with CD.

The primary objective of this study is to determine the effect of growth hormone (GH) therapy upon colon mucosal healing in a 12 week randomized trial in children with Crohn's Disease (CD). Children with active CD will be randomized to GH + prednisone (GP) or prednisone alone (P) for a 12 week period. This study also involves a 52 week extension phase where all participants that meet eligibility will be given the opportunity to take or continue taking growth hormone for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age ≥ 5 years.
* Diagnosis of Crohn's disease (CD) with ileo-colonic involvement as determined by standard clinical, radiological, and pathological criteria.
* Moderate to severely active CD as defined by a PCDAI (Pediatric Crohn's Disease Activity Index) ≥ 30.
* Currently taking Prednisone or Budesonide at starting dose (not tapering)
* May continue stable doses of AZA/6-MP, methotrexate, and/or mesalamine at entry.
* For the 52 week extension, baseline bone age ≤ 12 years for girls and ≤ 13 years for boys.
* For the 52 week extension phase, remission or mild Crohn's disease as determined by a PCDAI < 30.

Exclusion Criteria:

* Acute critical illness
* Active neoplasia
* Diabetes mellitus
* History of intracranial lesion and/or neoplasia
* Severe disease requiring hospitalization for treatment
* Current therapy with infliximab as this may independently rapidly reduce clinical disease activity and promote mucosal healing
* Use of prednisone or budesonide and in tapering phase
* Family history of colorectal cancer before age 50
* Personal or familial history of familial polyposis syndrome
* Pregnancy (positive pregnancy test) prior to randomization
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial other than the Pediatric IBD (Inflammatory Bowel Disease) registry

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-04; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Denson, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 98 subjects were assessed for eligibility, 76 did not meet inclusion criteria, 21 refused to participate
Pre-assignment Details: 21 subjects enrolled, one withdrew consent prior to randomization.
Groups:
- Growth Hormone Plus Corticosteroid (CTX): Growth Hormone (nutropin AQ 0.075 mg/kg/day subcutaneously daily)
- Corticosteroid (CTX): Subjects took corticosteroid as prescribed by their physician
Period: Baseline (0 Through 12 Weeks)
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Started | 10 (11 subjects allocated to Group A; one withdrew consent, only 10 receieved intervention.) | 10
Analyzed | 10 | 10
Completed | 10 | 9 (One subject discontinued intervention because of active disease requiring imfliximab)
Not Completed | 0 | 1
Period: Week 12 to Week 24
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Started | 10 | 9
Analyzed | 9 | 9
Completed | 9 (One subject withdrew consent) | 9 (one subject discontinued intervention due to active disease requiring surgery)
Not Completed | 1 | 0
Period: 52 Week Extension Phase
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Started | 9 | 8
Analyzed | 9 | 8
Completed | 5 (Extension phase ends when subjects discontinue intervention due to active disease or reaches week 64) | 3 (Extension phase ends when subjects discontinue intervention due to active disease or reaches week 64)
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Number; unit: participants]
  <=18 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (3) | 13 (3) | 13 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Crohn's Disease Histologic Index of Severity (CDHIS)
Description: The CDHIS was developed and validated in order to determine the effect of therapies upon histologic disease activity in Crohn's Disease. It has been used to assess mucosal healing in response to infliximab and 6-MP/AZA.It contains eight items which reflect epithelial injury, mucosal inflammation, and the extent of involvement. Scores range from 0-16, with patients with moderate to severely active CD typically having scores of 6-12. It was computed by a GI pathologist. The higher the score indicates worsening of disease, the lowest score is 0 and highest possible is 16
Time Frame: Baseline and 12 weeks
Measure: Number (95% Confidence Interval); unit: scores on a scale
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Number analyzed (Participants) | 10 | 10
scores on a scale
  Baseline | 7 [5 to 9] | 8 [6 to 10]
  Week 12 | 6 [4 to 8] | 8 [5 to 10]

2. Secondary Outcome: Serum IGF-1 (Insulin-like Growth Factor 1)z Score
Description: Elevated serum IGF-1 levels have been implicated in the development of colorectal cancer, both in the general population and in patients with an excess of growth hormone production. The serum IGF-1 levels were monitored to maintain them in the physiologic range during growth hormone therapy to reduce the risk of tumorigenesis.
  The levels are reported as a z score, a statistical way of standardizing data. The standard deviation is the unit of measurement of the z-score. Each z score corresponds to a point in a normal distribution, describing how much a point deviates from a mean.
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Error); unit: Z score
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Number analyzed (Participants) | 10 | 10
Z score
  Baseline | -0.4 (0.6) | -0.7 (0.3)
  Week 12 | 1.8 (1) | -1 (0.3)
  Week 24 | 3.3 (1.5) | 3.8 (1)

3. Secondary Outcome: IMPACT III Score
Description: Health-related quality of life (QOL)was assessed using the IMPACT 111 questionnnaire. It is a self-administered 35 item questionnaire which typically takes 10-15 minutes to complete. Scores range from 0-350, with higher scores reflecting better perceived quality of life.
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 134 [120 to 148] | 132 [119 to 146]
  Week 12 | 143 [129 to 157] | 136 [123 to 150]

4. Secondary Outcome: Pediatric Crohn's Disease Activity Index (PCDAI)
Description: The PCDAI is a previously validated measure of clinical disease activity for children with CD. It contains three self-report items which reflect patient abdominal pain, diarrhea, and general well being; three laboratory values; height and weight velocity; and three physical examination parameters reflecting abdominal tenderness, perirectal disease, and extra-intestinal manifestations. Scores may range from 0-100. Remission is defined as 0-10, mild disease as 10-30, and moderate to severe disease as greater than 30.
Time Frame: Baseline, 12 and 24 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 32 [20 to 43] | 33 [25 to 40]
  Week 12 | 8 [2 to 14] | 22 [14 to 30]
  Week 24 | 9 [2 to 14] | 6 [1 to 10]
Statistical Analysis 1: Comparison: Growth Hormone Plus Corticosteroid (CTX) vs Corticosteroid (CTX); Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = 14

5. Secondary Outcome: Total Corticosteroid Use
Description: The total corticosteroid use over 12 weeks between groups, using the unpaired t test.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: mg
Arm/Group | Growth Hormone Plus Cortecosteroid | Cortecosteroids Alone
Number analyzed (Participants) | 10 | 8
mg
  prednisone | 22 (8) | 28 (10)
  budesonide | 7 (4) | 8 (3)

6. Secondary Outcome: Crohn's Disease Endoscopic Index of Severity (CDEIS)
Description: Measure of mucosal disease at baseline and week 12 obtained during colonoscopy. The CDEIS score generally ranges from 0-30. A higher score indicates more severe mucosal inflammation.
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Baseline | 9 [-1 to 18] | 8 [2 to 13]
  Week 12 | 3 [1 to 6] | 6 [1 to 12]

7. Secondary Outcome: Height Velocity
Description: Height velocity was computed every 12 weeks up to week 64 and then yearly during the Maintenance study. Since 40 to 80% of children with Crohn's disease have significant growth failure at diagnosis, height velocity is used to track for changes in height.
  It is calculated by measuring height at two points of time and then dividing the change by the amount of time.
Time Frame: Baseline, week 12, 24 and 48
Measure: Mean (Standard Error); unit: cm/year
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Number analyzed (Participants) | 10 | 10
cm/year
  Baseline | 5 (1) | 3 (1)
  Week 12 | 8 (1) | 3 (1)
  Week 24 | 9 (1) | 7 (1)

8. Secondary Outcome: Fecal Calprotectin
Description: Fecal calprotectin is a previously validated stool marker of intestinal inflammation in Crohn's Disease.
Time Frame: At 24 and 64 weeks
Measure: Mean (95% Confidence Interval); unit: micrograms per gram (microg/g)
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX)
Number analyzed (Participants) | 10 | 10
micrograms per gram (microg/g)
  Baseline | 863 [517 to 1209] | 904 [540 to 1269]
  Week 12 | 868 [523 to 1214] | 656 [310 to 1002]

ADVERSE EVENTS:
Groups:
- Corticosteroid (CTX): Subjects took corticosteroid as recommended by their physician
- Extension Phase: Eligible subjects from both group A and group B continued on growth hormone in a 52 week extension phase
Arm/Group | Growth Hormone Plus Corticosteroid (CTX) | Corticosteroid (CTX) | Extension Phase
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 2/17
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone Plus Corticosteroid (CTX) (N=10) | Corticosteroid (CTX) (N=10) | Extension Phase (N=17)
Bruising at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Growth Hormone Plus Corticosteroid (CTX) (N=10) | Corticosteroid (CTX) (N=10) | Extension Phase (N=17)
Allergic Rhinitis (Immune system disorders) | 2 (2) | 0 (0) | 3 (3)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Lactose intolerant (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
ANC elevated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Basophils elevated (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased hematocrit (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophils elevated (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3)
Ferritin decrease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hematocrit decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Hematocrit elevated (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 1 (1)
Iron level decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Iron level elevated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Lymphocytes elevated (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Monocytes elevated (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 3 (4)
RBC decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
RBC elevated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
RDW elevated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Sedimentation Rate Elevated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Segs elevated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3)
Fever (General disorders) | 2 (3) | 2 (2) | 8 (8)
Increased thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Weight loss (General disorders) | 0 (0) | 1 (1) | 3 (3)
Bruising at injection site (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 5 (9)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Insect bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Seborrhea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fecal urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 6 (8)
Hemorrhage nasal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Colitis, infectious (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (5)
Oral thrush infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vaginal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ALT decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
ALT increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
AST increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (9)
Alkaline phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anion gap high (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anti-mitochondrial antibody (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
BUN (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
BUN decreased (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 2 (2)
BUN elevated (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Bilirubin increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bicarbonate elevated (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (6)
Blood glucose decreased (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
CRP elevated (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Chloride elevated (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2/10 (2)
Creatnine decreased (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 3 (3)
Creatinine elevated (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperinsulinemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Urine calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Concussion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 1 (3) | 1 (1) | 7 (7)
Back pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 4 (4) | 3 (3)
Joint Pain (General disorders) | 6 (6) | 1 (1) | 3 (3)
Myalgia (General disorders) | 0 (0) | 1 (1) | 2/10 (2)
Pain in extremity (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (General disorders) | 1 (1) | 2 (2) | 2 (2)
Rectal pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Shoulder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (General disorders) | 2 (2) | 4 (4) | 2 (2)
Sinus congestion (General disorders) | 0 (0) | 1 (3) | 1 (1)
Dysuria (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No